CLINICAL TRIAL: NCT03479177
Title: The Effect of a Home-Based High Intensity Interval Training Intervention on Increasing Exercise Among Low Active Adults
Brief Title: Home-Based High Intensity Interval Training Intervention for Low Active Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00001989
Record Dates: First submitted 2018-01-29; First posted 2018-03-27 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental): The exercise group will participate in a home and telephone-based program consisting of a 12-week high intensity interval training workout (HIIT). The home-based exercise sessions will be prescribed by the program exercise counselor, with a goal to exercise three times per week. The program will be tailored to meet specific fitness and strength needs of the participant. The participant will receive weekly telephone calls during the first month and bi-weekly calls during months 2 and 3. At 12 weeks, participants in both the exercise and wait-list control group will complete online questionnaires. The ActiGraph will be returned to the University of Minnesota research staff via a pre-paid postage envelope.
  Interventions: Behavioral: High Intensity Interval Training
- Wait-List Control Group (No Intervention): Participants in the wait-list control condition will have the option of receiving the exercise intervention program after completion of the final assessment.

INTERVENTIONS:
Behavioral: High Intensity Interval Training — The exercise sessions will be based on exercises the participant can confidentially engage in (regular push-ups vs. knee push-ups vs. wall push-ups). The goal will be to engage in three exercise sessions per week. The participants will receive weekly telephone calls during the first month and bi-weekly calls during months 2 and 3. The exercise counselor will also engage in dialogue that will motivate the participant to exercise.
  Arms: High Intensity Interval Training

SUMMARY:
The purpose of this study is to examine the effect of a home-based high intensity interval training intervention on exercise among low active adults (defined as engaging in exercise 90 minutes or less per week). Participants will be randomly assigned to a HIIT-based intervention or a wait-list control each lasting 12 weeks (participants in the wait-list control condition will have the option of receiving the HIIT intervention following the 12 weeks).

DETAILED DESCRIPTION:
The intervention will be a 12-week high intensity interval training workout that will consist of home-based exercise sessions prescribed by the exercise counselor. The exercise sessions will be based on exercises the participant can confidentially engage in (regular push-ups vs. knee push-ups vs. wall push-ups). The goal will be to engage in three exercise sessions per week. The participants will receive weekly telephone calls during the first month and bi-weekly calls during months 2 and 3. The exercise counselor will also engage in dialogue that will motivate the participant to exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Exercising for 90 minutes or less each week
* Access to the Internet

Exclusion Criteria:

* A history of coronary heart disease (history of myocardial infarction, symptoms of angina)
* Orthopedic problems that would limit physical activity participation
* Diabetes
* Stroke
* Osteoarthritis
* Any other medical condition that may make physical activity unsafe or unwise.
* Current or planned pregnancy
* Psychosis or current suicidal ideation
* Psychiatric hospitalization within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Exercise minutes per week | Change from Baseline to 12 weeks
  Exercise minutes per week as assessed by an accelerometer for one week at baseline and 12 weeks. Higher reported minutes per week indicates a higher level of physical activity.

SECONDARY OUTCOMES:
Biometrics | Change from Baseline to 12 weeks
  Body Mass Index will be calculated based on combining weight and height to report BMI as kg/m*2. The higher the number (level) of BMI, indicative of higher weight to height ratio.
Social Support for Exercise Questionnaire | Change from Baseline to 12 weeks
  Assesses the degree to which the individuals has friends and family who support their exercise. Participants rate how often family member or friend expresses social support for physical activity with scale (0=none, 4=very often). Overall total score range 0- 104 with subscales for family (0-52) and friends (0-52).
Physical Activity Self-efficacy Questionnaire | Change from Baseline to 12 weeks
  Assesses the amount of confidence the individual has to engage in exercise. Five questions, responses are on a scale from 1- 5 with participants indicating how confident they are on that scale of engaging in exercise in that situation (1=not at all confident, 5=extremely confident). Range of scores 5-25.
Physical Activity Enjoyment Scale (PACES) | Change from Baseline to 12 weeks
  Assesses the degree to which the individual enjoys exercise. The Physical Activity Enjoyment Scale is an 18-item scale that assesses enjoyment for physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" using a 7- point bipolar Likert scale, from 1 (I enjoy it) to 7 (I hate it). Eleven items were negatively worded and seven items were positively worded. After reverse scoring the 11negatively worded items, an overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible. Higher scores indicate higher enjoyment.
Outcome Expectancies Questionnaire | Change from Baseline to 12 weeks
  Assesses what benefits the individual expects to gain from exercise. Responses on a scale from 1-5 (1=strongly disagree, 5=strongly agree), with participants indicating how strongly they agree to potential outcomes of exercise. Scores range from 9-45 with higher scores indicating greater outcome expectation.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Lewis, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota- Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Lewis BA, Schuver K, Dunsiger S. Evaluating the feasibility and efficacy of a home-based combined high intensity interval and moderate intensity training program for increasing physical activity among low-active adults: A randomized pilot trial. PLoS One. 2023 Feb 21;18(2):e0281985. doi: 10.1371/journal.pone.0281985. eCollection 2023. PMID 36809292